CLINICAL TRIAL: NCT05696028
Title: Resident Doctor at Clinical Pathology Departement
Brief Title: Comparison of Different Gfr Measurements in Chronic Kidney Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa zidan, Resident doctor at clinical pathology departement, Assiut University
Other Study IDs: Clinical pathology
Record Dates: First submitted 2022-12-28; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Gamma counter — DTpA
  Other Names: Radionucide method

SUMMARY:
Comparison of different Gfr measurements in Chronic Kidney Diseases

DETAILED DESCRIPTION:
Comparison of gfr measured by different method as radionuclide method and creatinine clearance

ELIGIBILITY:
Inclusion Criteria:

* patients with proven or suspected CKD who will be referred to nuclear medicine departement of Assuit University hospital and will undergo dynamic renal imaging.

Exclusion Criteria:

* Severely ill patients
* Disturbed conscious level
* Patients on dialysis
* patients have oedema or ascites

Ages: 40 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients proven or suspected CKD
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Is to Compare gfr measured by radionuclide method to gfr measured by creatinine clearance in patients with CKD | 1year
  Gfr can be measured by quantification of plasma and standard volume sample using a quality controlled gamma_counter and Gamma camera these techniques the central assumption that the tracer is cleared solely by glomerular filtration.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Zidan, doctor, Principal Investigator — Assiut University